CLINICAL TRIAL: NCT01461018
Title: A Multicenter Study of Long-Term Clinical Outcomes of Immune Globulin Subcutaneous (Human) (SCIG) IgPro20 in Subjects With Primary Immunodeficiency
Brief Title: Multicenter Study of Long-Term Clinical Outcomes of Subcutaneous Immune Globulin IgPro20 in Subjects With Primary Immunodeficiency (Japan Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IgPro20_3006
Record Dates: First submitted 2011-10-24; First posted 2011-10-27 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Primary Immune Deficiency
Keywords: Immune globulin subcutaneous; SCIG; Primary immunodeficiency; PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Hizentra

ARMS (1):
- IgPro20 (Experimental)
  Interventions: Biological: Immune globulin subcutaneous (Human)

INTERVENTIONS:
Biological: Immune globulin subcutaneous (Human) — IgPro20 is a 20% (weight per volume [w/v]) liquid formulation of human immunoglobulin for subcutaneous (SC) use.
  Other Names: Hizentra

SUMMARY:
The purpose of this study is to assess the long-term efficacy, tolerability, and safety of IgPro20 in subjects with primary immunodeficiency (PID) as an extension to the preceding follow-up study ZLB07_001CR (NCT01458171).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the preceding follow-up study ZLB07_001CR.
* Written informed consent by the subject/parent/legally acceptable representative. Written assent for an underage subject (≥7 years and <20 years of age at the time of obtaining informed consent), according to the competencies of the subject.

Exclusion Criteria:

* Pregnancy or nursing mother.
* Participation in a study with an investigational medicinal product (IMP) within 3 months prior to enrollment except for study ZLB07_001CR.
* Subjects who are planning to donate blood during the study.
* Known or suspected antibodies to the IMP, or to excipients of the IMP.
* Treatment with another immunoglobulin G (IgG) within 3 months prior to the study.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Annualized rate of infection episodes | Up to 36 months

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs) | Up to 36 months
Percentage of subjects with adverse events (AEs) | Up to 36 months
Rate of AEs per infusion | Up to 36 months
Annualized rate of clinically documented serious bacterial infections (SBIs) | Up to 36 months
  SBIs are defined as bacterial pneumonia, bacteremia and septicemia, osteomyelitis/septic arthritis, bacterial meningitis, or visceral abscess.
Number of days out of work/school/kindergarten/day care or unable to perform normal daily activities due to infections | Up to 36 months
Number of days of hospitalization due to infections | Up to 36 months
Duration of use of antibiotics for infection prophylaxis and treatment | Up to 36 months
Median serum IgG concentration | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Yusuke Watanabe, Study Director — CSL Behring K.K.
Locations (9):
- Japan (9):
  - Study site, Nagoya, Aichi Pref.
  - Study site, Chiba, Chiba Pref.
  - Study site, Fukuoka, Fukuoka
  - Study site, Gifu, Gifu Pref.
  - Study Site, Sapporo, Hokkaido
  - Study site, Moriguchi, Osaka
  - Study site, Koshigaya, Saitama Pref.
  - Study site, Tokorozawa, Saitama Pref.
  - Study site, Bunkyō City, Tokyo Metropolitan